CLINICAL TRIAL: NCT04172207
Title: Effects of Antibiotic Consumption Time on Gingival-biopsy and Oral-smear Samples.
Brief Title: Antibiotic, Gingival-biopsy, and Oral-smear Samples.
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Begum Alkan, Principal Investigator, Istanbul Medipol University Hospital
Other Study IDs: Istanbul Medipol University
Record Dates: First submitted 2019-11-08; First posted 2019-11-21 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Anti-bacterial Agents; Chromosome-defective Micronuclei; Cytology; Histopathology
MeSH Terms: conditions — Micronuclei, Chromosome-Defective

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Results of study groups.
  Interventions: Other: Sampling

INTERVENTIONS:
Other: Sampling — After periodontal parameters measured, smear samples were obtained from the buccal mucosa and keratinized gingiva, and then a gingival biopsy was performed from the upper premolars.

SUMMARY:
Antimicrobial or antibiotic agents, which are essential to prevent and treat bacterial infectious diseases, have become one of the most widely used drugs in the world. In the European region, the highest rates of antibiotic consumption are reported in Turkey. There is a nearly fivefold difference between Turkey and the lowest consuming countries.

Studies in dentistry evaluate participants according to the basis of predefined criteria. History of antibiotic consumption is one of the most common exclusion criteria for periodontal trials. However, there is still disagreement on how long the effect of systemic antibiotic agents on the oral mucosa and periodontal tissue lasts. It is unclear whether the timing of antibiotic consumption should be an exclusion criterion for genetic damage and histological studies during the selection of healthy participants.

Periodontal status of participants in study groups is described as with or without periodontitis in many studies, because of the lack of clear definitions of periodontal health and gingivitis. It should be recognized that even the lack of visual signs of inflammation, some mild histopathological changes can be seen in the periodontium. Consequently, for the real diagnosis of the clinically healthy periodontium, clinical findings should be supported and confirmed with histological results.

Micronuclei (Mn) are observed as abnormal nuclear structures and indicators of chromosomal level DNA damage. The oral mucosa epithelium is an immunologic barrier and affected by chemical factors such as antibiotic consumption. The Mn test to exfoliated epithelial cells from the oral cavity is utilized as a non-invasive diagnostic technique for monitoring the status of oral health. To our knowledge, no studies have been conducted on the comparison of the impacts of the timing of antibiotic consumption on human periodontal tissues and oral smear samples. The present study is undertaken to determine whether the different timing of antibiotic (amoxicillin) therapy has effects on the histopathology of gingiva and genetic damage of exfoliated cells from oral mucosa in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Systemically and periodontally healthy participants
* Presence of probing depth (PD) of ≤ 3 mm14 and bleeding on probing (BOP) ˂ 10%15
* No clinical evidence of gingival recession (GR), clinic attachment loss or radiographic evidence of alveolar bone loss
* No periodontal treatment within the last 12 months

Exclusion Criteria:

* Smoking, alcohol or drug abuse
* Any systemic condition would affect the periodontal health (i.e., pregnancy, lactation, ovulation, and diabetes mellitus)
* A history of contagious disease
* Periodontal treatment within the last 12 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 45 systemically and periodontally healthy participants, who were referred to the clinics of the Department of Periodontology, Faculty of Dentistry, Istanbul Medipol University between 2018 and 2019 for routine periodontal visits, were included in this study. Participants were divided into three groups based on the history of oral antibiotic (1 g amoxicillin bid, two times a day) consumption for upper respiratory tract infection in the previous 12 months: group I (n = 19), participants used antibiotic between 12-6 months before the sampling; group II (n = 13), participants used antibiotic between 6-3 months before the sampling; group III (n = 13), participants used antibiotic within a period of 1-month before to sampling.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Effects of antibiotics on gingiva confirmed by histopathology. | 1-week
  Modified histological criteria was the measurement used for the semi-quantitative histological assessment of gingival damage. Cellular components, vascularization, cell infiltration, necrosis, pyknotic nucleus, hyperemia, fibrosis, ulceration, atrophy, apoptosis, and rete peg configuration were scored by using a scale ranging from 0 to 3 (none : 0, mild: 1, moderate: 2, and severe : 3) for each criterion.
Effects of antibiotics on buccal and oral smear confirmed by quantitative determination of the micronuclei. | 1-week
  The method has been applied both for monitoring chromosome damage and/or proteins may also result in unsuccessful attachment of a whole chromosome at anaphase stage which subsequently also gives rise to a micronucleus. Thus, quantitative determination of the micronuclei are unique amongst cytogenetic tests in that it provides a reliable measure of both chromosome loss and breakage.

CONTACTS AND LOCATIONS:
Locations (1):
- Begum Alkan, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No